CLINICAL TRIAL: NCT03014427
Title: Development of a Biological Database in the Field of Operative Intensive Care for the Recording of Clinically Relevant Parameters of Critically Ill Intensive Patients
Brief Title: Development of a Biological Database in the Field of Operative Intensive Care
Acronym: Biobank OIM
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-151
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Intensive Care in General

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples With DNA — Patients can give consent to the analysis of DNA seperately.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biological Database — Biological Database

SUMMARY:
The storage and use of biomaterial samples is an important requirement for accompanying research and the acquisition of new knowledge to improve prognosis and therapy. Biobanking is explicitly recommended in official guidelines. In order to preserve the biomaterial, the patient must consent to the removal, transfer and storage of the biomaterial separately from the consent to the register. The biomaterial is taken at times at which a blood or urine sampling takes place anyway in the clinical routine. Therefore no additional interventions are necessary.

DETAILED DESCRIPTION:
The storage and use of biomaterial samples is an important requirement for accompanying research and the acquisition of new knowledge to improve prognosis and therapy. Biobanking is explicitly recommended in official guidelines. In order to preserve the biomaterial, the patient must consent to the removal, transfer and storage of the biomaterial separately from the consent to the register. The biomaterial is taken at times at which a blood or urine sampling takes place anyway in the clinical routine. Therefore no additional interventions are necessary.

Sample volumes are defined as follows:

* Peripheral blood: up to a total of 150 ml distributed to a maximum of 10 morning blood samples (approximately 15 ml blood per blood sample) during the inpatient stay in the intensive care unit (fixed times are admission and discharge of the intensive care unit)
* Urine: a total of up to 200 ml of catheter urine distributed to a maximum of 10 morning withdrawals during inpatient stays in the intensive care unit (defined times are admission and discharge from the intensive care unit)

ELIGIBILITY:
Inclusion Criteria:

* patients after admission to the intensive care unit
* 18 years or older
* signed informed consent

Exclusion Criteria:

* No exclusion criteria are formulated with regard to the objective of the register to record intensive care patients in general. Patients with multiple comorbidities, organ dysfunctions, and non-compliance for a curatively-intended therapy should also be recorded in the register. A palliative treatment or decision for best supportive care is not an exclusion criterion for registering.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients in general
Sampling Method: Non-Probability Sample
Enrollment: 99999999 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2050-02 (Estimated); Study Completion 2050-02 (Estimated)

PRIMARY OUTCOMES:
Interleukin 6 value [nmol/l] | 10 days
  Record of clinically relevant parameters
Interleukin 10 [nmol/l] | 10 days
  Record of clinically relevant parameters
Adrenomedullin value [nmol/l] | 10 days
  Record of clinically relevant parameters
Tumornekrosefaktor alpha [nmol/l] | 10 days
  Record of clinically relevant parameters
Procalcitonin [nmol/l] | 10 days
  Record of clinically relevant parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stoppe, Dr. med., Principal Investigator — Operative Medicine and Intensive Care, RWTH Aachen University
Locations (1):
- Uniklinik RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bestehorn K. [Medical registries]. Med Klin (Munich). 2005 Nov 15;100(11):722-8. doi: 10.1007/s00063-005-1098-x. German. PMID 16328180
- [Background] Schott G, Berthold HK. Pharmakovigilanz: Empfehlungen zur Meldung unerwünschter Arzneimittelwirkungen durch die Ärzteschaft. Arzneiverordnung in der Praxis. 2005.